CLINICAL TRIAL: NCT04087486
Title: Validation of an Ecological Organization and Problem Solving Test (TEM-PRO)
Brief Title: Validation of an Ecological Organization and Problem Solving Test (TEM-PRO) in Vocational Rehabilitation
Acronym: TEM-PRO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Other Study IDs: CliniqueRR-07
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Multiple errands tests
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Implementation of a behavioural test for patients with TBI — The following data will be collected: (1) sociodemographic variables (2); clinical and psychological data; (3) functional tests (neuropsychological testing, TEM version CRR and TEM-PRO).
  On day one, patients will undergo standard neuropsychological tests and questionnaires listed hereafter, which are commonly used in the clinical practice at the CRR.
  * The Patient Competency Rating Scale (PCRS)
  * TEM (Multiple errands test)
  * GREFEX
  * 5 POINTS TEST
  * TAP 2.3
  * Behavioral Assessment of the Dysexecutives Syndrome (BADS)
  On day two, the patients will perform the TEM-PRO test ambulatory in our vocation rehabilitation unit.
  "Predictors" variables will be collected before testing: Sociodemographic: age, sex, education, marital status, mother language, time since TBI, severity of the TBI (moderate or severe), type of lesion (contusion, diffuse axonal injury grade 1-3, ischemic or other complications), history of TBI, stroke or meningitis.

SUMMARY:
Standard neuropsychological evaluations after severe TBI (traumatic brain injury) often minimizes the executive deficits, these latter are known to seriously impair return to work. Therefore, we developed an ecological organization and problem-solving test in a vocational setting called the TEM-PRO. The test consists of 4 activities of variable complexity, collection and redaction of information and demands to follow well defined rules.

DETAILED DESCRIPTION:
While there may be many reasons for obtaining neuropsychological assessement after TBI, predication of the real world functioning is generally the final goal. Among the cognitive deficits, the dysexecutive syndrome is certainly the most disabling in impeding to return to work. The classical neuropsychological tests often fail to asses theses deficits adequately. Several more ecological tests have been previously developed. Based on the multiple errands test and the six elements test, we built up first an ecological test over 60 minutes for activities of the daily living (test des errances multiples, " TEM, version CRR "). Used regularly in the clinical setting, it was able to evaluate the functional aptitudes of the patients and was useful to complete the classical neuropsychological tests. However test duration is too short and activities are far away from real work scenarios to test working aptitudes. Therefore we developed a new executive-ecological test in a vocational setting (TEM-PRO). The adaptation of the original test in a vocational setting induces the addition of 4 activities of variable complexity, research and redaction of information and demands to follow well defined rules. Skills that are solicited are planning, selective and sustained attention, prospective memory, organization, problems solving and behavior adaption over a long period of time. Based on a pilot study with patients without neurological deficit we assessed that our test displayed good sensitivity without ceiling effect. It allowed a quantitative and differentiated evaluation, a classification of various error types (interpretation and judgment failure, rule breaks, task failures and inefficiencies) and provided a qualitative behavioral analysis.

ELIGIBILITY:
Inclusion Criteria:

French speaking patients, older than 18 years, able to understand and sign the study informed consent, able to answer questionnaires used in the study, suffering from moderate to severe TBI, without invalidate psychiatric comorbidities, without severe memory impairment, capable to participate for 4h in a vocational activity, planning to return to work. Patients still receiving compensation and patients returned to work will be included

Exclusion Criteria:

alcohol or drug abuse, severe physical disability interfering with the test (modified Ranking score >1), under legal custody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a moderate to severe traumatic brain injury returning to work
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the feasibility of the test. | 2020
  Is it suitable for TBI patients?

SECONDARY OUTCOMES:
Evaluation of the criterion validity of the TEM-PRO | 2020
  Evaluation of the reproducibility of the test
Comparaison of the diagnostic value of the TEM-PRO with the classical Neuropsychological test and the TEM. | 2020
  Comparison with existing tests
Evaluation of the association between RTW and TEM-PRO | 2022
  Can the test be a predictor of RTW?

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Mühl, MD, Principal Investigator — Clinique romande de réadaptation
Locations (1):
- Clinique romande de réadaptation, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided